CLINICAL TRIAL: NCT02847559
Title: A Phase 2, Single Arm, Multi-center, Open Label Trial Combining Optune With Concurrent Bevacizumab in the Setting of Recurrent or Progressive Meningioma
Brief Title: Optune Delivered Electric Field Therapy and Bevacizumab in Treating Patients With Recurrent or Progressive Grade 2 or 3 Meningioma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: NovoCure Ltd. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 16C02; STU00203030 (CTRP (Clinical Trial Reporting Program)); NU 16C02 (Other: Northwestern University); P30CA060553 (NIH); NCI-2016-01026 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Anaplastic (Malignant) Meningioma; Atypical Meningioma; Grade II Meningioma; Grade III Meningioma; Recurrent Meningioma; Supratentorial Meningioma
MeSH Terms: conditions — Meningioma | interventions — Bevacizumab; Immunoglobulin G; Disulfides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (1):
- Treatment (bevacizumab, electric field therapy) (Experimental): Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15 of courses 1-4. Beginning on day 1 of course 5, patients may choose to receive bevacizumab IV every 3 weeks or remain on the every 2-week schedule. Patients also undergo electric field therapy using Optune (formerly NovoTTF-200A System) daily over 18 hours. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Procedure: Electric Field Therapy; Device: NovoTTF-200A Device; Procedure: Quality-of-Life Assessment

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
Procedure: Electric Field Therapy — Undergo electric field therapy using Optune device
Device: NovoTTF-200A Device — Undergo electric field therapy using Optune device
  Other Names: NovoTTF-200A; NovoTTF-200A System; NovoTTFields; NovoTumor Treatment Fields; Optune; Optune Device
Procedure: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
The purpose of this research study is to determine the effects bevacizumab (the study drug) combined with Optune (the study device) tumor treatment field therapy has on meningiomas. Bevacizumab is considered investigational because the US Food and Drug Administration (FDA) has not approved its use for the treatment of meningiomas. The study drug is a medication that blocks the growth of new blood vessels. It is thought that the study drug may interfere with the growth of new blood vessels and therefore might stop tumor growth, and possibly shrink the tumor by keeping it from receiving nutrients and oxygen supplied by the blood vessels. Optune is also considered investigational because the US FDA has not approved its use for the treatment of meningiomas. Optune is a device that the patient will wear and use for at least 18 hours of each day. It delivers alternating electrical current to the patient's brain tumor and by doing so interrupts a process called mitosis. Mitosis needs to occur in order for cell division to occur and allows tumors to grow. By slowing this process, we hypothesize that meningioma growth may also be slowed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine progression free survival (PFS) for 6 months (PFS-6) in patients with recurrent or progressive meningioma.

SECONDARY OBJECTIVES:

I. To determine overall survival (OS). II. To determine tumor response rate (TRR). III. To assess quality of life with treatment (QOL) using Functional Assessment of Cancer Therapy-Brain (FACT-Br) questionnaire.

OUTLINE:

Patients receive bevacizumab intravenously (IV) over 30-90 minutes on days 1 and 15 of courses 1-4. Beginning on day 1 of course 5, patients may choose to receive bevacizumab IV every 3 weeks or remain on the every 2-week schedule. Patients also undergo electric field therapy using Optune (formerly NovoTTF-200A System) daily over 18 hours. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologic diagnosis of meningioma, World Health Organization (WHO) grade 2 or 3 (atypical or anaplastic)
* Patient's tumor must have a supratentorial component
* Patients must have measurable or non-measurable (evaluable) disease recurrence; recurrence must be documented by magnetic resonance imaging (MRI) or computed tomography (CT) scan
* All patients must have developed recurrent disease/progression (evidence of recurrence to be established by MRI or CT scan with contrast; there is no limit to the number of relapses) after receiving all standard treatments, which must include the following:

  * Surgical resection, if possible;
  * Definitive radiation therapy for unresectable meningioma, or for recurrent meningioma after resection (Note: At registration, patients must be at least 28 days post-surgery, and must be at least 28 days post-radiation therapy, with resolution of related cytotoxicities down to grade 2)
* Patients may have had previous systemic treatment regimens with the exception of bevacizumab (no limit to number of prior therapies); a 4 week wash-out period prior to registration is mandatory for all systemic treatments
* Life expectancy of at least 12 weeks
* Karnofsky performance status >= 60%
* Patients must have adequate bone marrow, kidney, and liver function, (within 14 days prior to registration), defined as:
* Absolute neutrophil count (ANC) >= 1500/uL (with/without growth factor)
* Hemoglobin (Hgb) >= 9 g/dL (with/without transfusion)
* Platelets >= 100,000/L
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x institutional upper limit of normal (ULN)
* Total bilirubin =< 1.5 x institutional ULN
* Serum creatinine =< 1.5 x institutional ULN
* Females of child-bearing potential (FOCBP) and males with partners of childbearing potential must agree to use adequate contraception prior to study entry and for the duration of study treatment; should a female patient become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; likewise, if the female partner of a male patient becomes pregnant or suspect she is pregnant, he should inform his treating physician immediately

NOTE: A FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy
* Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)

  * FOCBP must have a negative serum or urine pregnancy test within 14 days prior to registration on study
  * Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study
  * Patients must be able to comply with all protocol requirements

Exclusion Criteria:

* Patients who have had major surgery or significant traumatic injury within 4 weeks prior to registration, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia), or patients that may require major surgery during the course of the study
* Patients who have had minor surgical procedures (with the exception of the placement of porta cath or other central venous access) within 7 days prior to registration
* Patients with infratentorial disease and spinal disease
* Patients may not be receiving any other investigational agents; (i.e. 28-day washout period from prior investigational drug is required)
* Patients may not receive any other anti-cancer therapies, within 28 days prior to registration and throughout the duration of this trial
* Previous treatment with bevacizumab
* Patients who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to bevacizumab are not eligible
* Patients with active implanted medical device, a skull defect (such as, missing bone with no replacement), a shunt or bullet fragments; examples of active electronic devices include deep brain stimulators, spinal cord stimulators, vagus nerve stimulators, pacemakers, defibrillators, and programmable shunts
* Patients with known sensitivity to conductive hydrogels like the gel used on electrocardiogram (ECG) stickers or transcutaneous electrical nerve stimulation (TENS) electrodes
* Patients with proteinuria within 14 days of registration as demonstrated by either: urine protein creatinine (UPC) ratio >= 1.0 at screening OR urine dipstick for proteinuria 2+ (patients discovered to have 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection, and must demonstrate =< 1 g of protein/24 hours to be eligible)
* Patients with a serious non-healing wound, active ulcer, or untreated bone fracture
* Patients with evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Patients with history of hematemesis or hemoptysis (defined as having bright red blood of 1/2 teaspoon or more per episode) within 28 days prior to registration
* History of myocardial infarction or unstable angina within 6 months of registration
* Inadequately controlled hypertension (defined as systolic blood pressure > 150 mmHg and /or diastolic blood pressure > 100 mmHg)
* History of stroke or transient ischemic attack within 6 months prior to registration
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to registration
* Chronic, systemic treatment with immunosuppressive agents; patients who require a stable dose of corticosteroids for control of cerebral edema are eligible; topical or inhaled steroids are also allowed
* Patients who have any severe and/or uncontrolled intercurrent medical conditions including, but not limited to any of the following, are not eligible:

  * Ongoing or active wound infection requiring concurrent systemic antibiotic treatment; there is no mandatory duration of time that a patient has to be off antibiotics, but the treating physician has to deem the infection as effectively treated prior to enrollment
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia (New York Heart Association [NYHA] criteria)
  * Psychiatric illness/social situations that would limit compliance with study requirements, prevent patient comprehension of the nature of, and risk associated with, the study
  * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints
* Female patients who are pregnant or nursing are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival for 6 months (PFS-6) | At 6 months
  Determine the efficacy of combination therapy of bevacizumab and Optune (TTF) as assessed by Progression Free Survival at 6 months

SECONDARY OUTCOMES:
Overall Survival (OS) | From time of registration to death, assessed up to 2 years
  OS will be defined from the time of registration to death and will be assessed for up to 2 years.
Tumor Response Rate (TRR) | At baseline and every eight weeks, assessed up to 12 months
  Imaging (MRI or CT scan) will assess radiographic response in terms of complete response, partial response, stable disease, and progressive disease. The iRANO criteria will be used for response assessment.
Quality of Life (QOL) with treatment using FACT-Br questionnaire | At baseline, on Day 1 of every cycle, and 1 month after the last dose of study drug
  To assess QOL with treatment the Functional Assessment of Cancer Therapy-Brain version 4.0 (FACT-Br) questionnaire will be administered.

CONTACTS AND LOCATIONS:
Overall Officials: Priya Kumthekar, MD, Principal Investigator — Northwestern University
Locations (8):
- United States (8):
  - John Wayne Cancer Center at Providence St. John's Health Center, Santa Monica, California
  - Miami Cancer Institute, Miami, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Northwestern University- Lake Forest Hospital, Lake Forest, Illinois
  - Northwestern Medicine/ Cadence Health - CDH, Winfield, Illinois
  - Vidant Medical Center, East Caroling University, Greenville, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No